CLINICAL TRIAL: NCT04641988
Title: Cardiac Biomarkers and Mortality in Critically Ill Patients With SARS-CoV-2 (COVID-19) : COROBIOCHIC
Brief Title: Cardiac Biomarkers and Mortality in Critically Ill Patients With SARS-CoV-2 (COVID-19)
Acronym: COROBIOCHIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0625
Record Dates: First submitted 2020-11-23; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Troponin; hs-cTnT; NT-proBNP
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To assess the prognostic value of high-sensitive cardiac troponin T (hs-cTnT) and N-terminal pro brain natriuretic peptide (NT-proBNP) at ICU admission in patients with coronavirus disease 2019 (COVID-19).

Design: Multicenter retrospective observational cohort study Setting: Three ICUs at three hospitals in Occitanie, France. Patients: Adults (≥ 18 years old) with laboratory-confirmed COVID-19 and at least one hs-cTnT measurement at ICU admission, from March 9, 2020, to May 9, 2020.

ELIGIBILITY:
Inclusion criteria:

- Adults (≥ 18 years old) with laboratory-confirmed COVID-19 and at least one hs-cTnT measurement at ICU admission

Exclusion criteria:

- Age < 18, pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
hs-cTnT | at ICU admission
  hs-cTnT

SECONDARY OUTCOMES:
NT-proBNP | at ICU admission
  NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: Romaric Larcher, MD, PharmD, MSc, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC